CLINICAL TRIAL: NCT01449526
Title: A Study to Evaluate the Safety and Efficacy of a New Silicone Hydrogel Contact Lens Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 661
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Myopia
Keywords: contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B&L Investigational Contact Lens (Experimental): The Bausch + Lomb investigational silicone hydrogel contact lens
  Interventions: Device: B&L Investigational Contact Lens
- B&L PureVision Contact Lens (Active Comparator): The Bausch + Lomb PureVision silicone hydrogel contact lens
  Interventions: Device: B&L PureVision Contact Lens

INTERVENTIONS:
Device: B&L Investigational Contact Lens — Lenses will be worn on a daily wear basis for 3 months, new lenses dispensed monthly.
  Arms: B&L Investigational Contact Lens
Device: B&L PureVision Contact Lens — Lenses will be worn on a daily wear basis for 3 months, new lenses dispensed monthly.
  Arms: B&L PureVision Contact Lens

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a new silicone hydrogel contact lens compared to the Bausch + Lomb PureVision contact lens when worn by adapted soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be myopic, and wear contact lenses in each eye.
* Subjects must be adapted soft contact lens wearers and agree to wear their study lenses on a daily wear basis for approximately 3 months.

Exclusion Criteria:

* Subjects who are older than age 40 on the date the informed consent (ICF) is signed.
* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects with any grade 2 or greater finding during the slit lamp examination.
* Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects who are allergic to any component in the study care products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a three month study enrolling 166 participants from 12 investigative sites in the United States. First participant was enroled on 08/08/2011, and last participant exited the study on 12/08/2011.
Pre-assignment Details: 166 participants were enrolled in the study with 158 participants completing the study. A minimum of 68 participants were to be of Japanese descent (both maternal and paternal grandparents born in Japan) for submission to the Japanese Regulatory Agency.
Period: Overall Study
Arm/Group | B&L Investigational Contact Lens | B&L PureVision Contact Lens
Started | 83 | 83
Completed | 81 | 77
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Symptoms/complaints | 0 | 1
Not completed — Lack of Motivation | 0 | 1
Not completed — Cannot maintain visits | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Eligible, Dispensed Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | B&L Investigational Contact Lens | B&L PureVision Contact Lens | Total
Number analyzed (Participants) | 83 | 83 | 166
Age, Continuous [Median (Full Range); unit: years] | 29.0 [19 to 40] | 29.0 [18 to 40] | 29.0 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 50 | 108
  Male | 25 | 33 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 53 | 55 | 108
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 2 | 2 | 4
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 83 | 166

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: Mean high contrast, distance logMAR VA for each eye between the Test and Control lenses. This measure is an average from 4 visits taking place over 3 months.
Time Frame: 4 visits over 3 months
Population: All Eligible, Dispensed Eyes
Measure: Least Squares Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | B&L Investigational Contact Lens | B&L PureVision Contact Lens
Number analyzed (Participants) | 83 | 83
Number analyzed (Eyes) | 166 | 166
LogMAR | -0.033 (0.054) | -0.038 (0.054)

2. Secondary Outcome: Slit Lamp > Grade 2
Description: Proportion of eyes with any slit lamp findings greater than grade 2 at any visit between the Test and Control lenses.
Time Frame: 3 months
Population: Number of dispensed eyes with non-missing scores in each treatment group.
Measure: Number; unit: eyes (2 per participant)
Units Other Than Participants: Eyes
Arm/Group | B&L Investigational Contact Lens | B&L PureVision Contact Lens
Number analyzed (Participants) | 82 | 82
Number analyzed (Eyes) | 164 | 164
eyes (2 per participant) | 2 | 5

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | B&L Investigational Contact Lens | B&L PureVision Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other